CLINICAL TRIAL: NCT03344211
Title: Immune Activation and Cellular Response From Enzalutamide Alone or With Radium223 in Men With Metastatic, Castration-Resistant Prostate Cancer
Brief Title: Enzalutamide With or Without Radium Ra 223 Dichloride in Patients With Metastatic, Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4P-16-2; NCI-2017-01418 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-16-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-11-04; First posted 2017-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Castration-Resistant Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (enzalutamide, radium 223) (Experimental): Patients receive enzalutamide PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive radium Ra 223 dichloride IV on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Radiation: Radium Ra 223 Dichloride
- Arm II (enzalutamide) (Experimental): Patients receive enzalutamide as in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM CHLORIDE RA-223; Radium-223 Dichloride; Xofigo
  Arms: Arm I (enzalutamide, radium 223)

SUMMARY:
This randomized phase II trial studies how well enzalutamide with or without radium Ra 223 dichloride in treating patients with castration-resistant prostate cancer that has spread to other places in the body. Enzalutamide is an androgen receptor inhibitor that may slow down the growth of prostate cancer by blocking the action of the male hormone testosterone and other male hormones called androgens. Radiation therapy uses high energy alpha particles to kill tumor cells and shrink tumors. Enzalutamide with or without radium Ra 223 dichloride may work better in treating patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate changes in prostate cancer bone involvement induced by enzalutamide alone or in combination with radium Ra 223 dichloride (radium 223), specifically extent of prostate cancer infiltration, androgen receptor (AR) signaling and hormone levels, hematopoietic composition, apoptosis and proliferation.

II. To evaluate the immune activation of enzalutamide alone, or with radium 223.

SECONDARY OBJECTIVES:

I. To describe the adverse event profile for the combination in this patient population.

II. Rate of undetectable prostate specific antigen (PSA) nadir, PSA and alkaline phosphatase changes, rate of symptomatic skeletal events at 12 months, and rate of PSA and radiographic progression at 12 months.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive enzalutamide orally (PO) daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive radium Ra 223 dichloride intravenously (IV) on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive enzalutamide as in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Men with metastatic, castration resistant prostate cancer involving the bone, which is symptomatic or asymptomatic
* Castration resistance will be defined as the development of disease progression, defined as one of the following:

  * Rising PSA x 2 values >= 2 weeks apart; minimum absolute PSA value 2 ng/mL
  * Radiographic progression, with at least 1 new site of metastasis
  * Symptomatic progression (ex: increase in pain despite stable imaging) AND despite ongoing luteinizing hormone-releasing hormone (LHRH) therapy OR testosterone level < 50
* Men must have osseous metastases, but the presence of visceral metastases will not exclude patients from participation

  * Prior external beam radiation therapy (> 4 weeks prior to enrollment) for palliation of osseous metastatic disease is allowed, provided there is at least one osseous metastasis which has not been irradiated and which can be biopsied
* No prior docetaxel or cabazitaxel chemotherapy for metastatic castration-resistant prostate cancer (mCRPC) (men treated with prior docetaxel administered as up-front therapy with androgen deprivation therapy [ADT] > 6 months ago will be eligible); prior abiraterone is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 9.5 g/dL
* Absolute neutrophil count >= 1,500
* Platelets >= 100,000
* Total bilirubin within normal institutional limits
* Creatinine clearance (calculated or measured) > 30 mL/min
* At least one risk factor predicting higher likelihood of bone marrow sample yield: elevated alkaline phosphatase, low hemoglobin, or elevated lactate dehydrogenase (LDH)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Prior treatment with docetaxel or cabazitaxel for mCRPC
* Prior treatment with ARN-509 or enzalutamide (there is a grace period for men who wish to enroll and who have recently started enzalutamide for the first time but have taken less than 15 days of therapy)

  * Concurrent use of androgen deprivation therapy aside from LHRH agonist or antagonist (i.e. bicalutamide, flutamide, nilutamide, abiraterone, ketoconazole, estrogen); there will be a 2 week wash-out period from the last dose of any of these agents until the first dose of enzalutamide on study; patients who have just started enzalutamide for fewer than 5 doses prior to enrollment in the trial are still considered eligible and not subject to wash-out
* Concurrent oral corticosteroid use aside from adrenal replacement, or use of other immunosuppressive agents (ex: infliximab); topical or inhaled steroids will be allowed
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium- 153, rhenium-186, or rhenium-188, or radium Ra 223 dichloride) for the treatment of bony metastases
* History of seizures except for remote with specific etiology which has resolved (ex: alcohol induced seizure); transient ischemic attack (TIA) or cerebrovascular accident (CVA) within last 6 months
* Known untreated central nervous system (CNS) metastases; leptomeningeal disease will be an absolute exclusion criterion due to limited life expectancy
* Chronic diarrhea > grade 1, or a diagnosis of Crohn?s or ulcerative colitis
* Known hepatitis (hep) B or C, or known cirrhosis (screening for viral hepatitis is not required)
* Uncontrolled intercurrent illness such as infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness which would limit compliance with study requirements
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI); treatment should be completed for spinal cord compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Changes in prostate cancer bone involvement | Up to 1.5 years
  Will be determined by standard pathologic analysis of the biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: David I Quinn, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California